CLINICAL TRIAL: NCT05866055
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled, Single- and Multiple-dose Escalation Study Evaluating the Safety, Pharmacokinetics, and Pharmacodynamics of VX-973 in Healthy Adults
Brief Title: A Phase 1 Dose Escalation Study of VX-973 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VX22-973-001; 2022-003301-30 (EudraCT Number)
Record Dates: First submitted 2023-04-24; First posted 2023-05-19 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part A: Single Ascending Dose (Experimental): Participants will be randomized to receive a single dose of VX-973 under fasted conditions.
  Interventions: Drug: VX-973
- Part B: Multiple Ascending Dose (Experimental): Participants will be randomized to receive multiple doses of VX-973 under fasted conditions. The dose and frequency will be determined based on Part A. Midazolam is planned to be administered as single oral doses of 2 mg first alone on Day -1 and then co-administered with study drug on Day 27.
  Interventions: Drug: VX-973; Drug: Midazolam
- Placebo Part A (Placebo Comparator): Participants will be randomized to receive placebo matched to VX-973.
  Interventions: Drug: Placebo
- Placebo Part B (Placebo Comparator): Participants will be randomized to receive placebo matched to VX-973. Midazolam is planned to be administered as single oral doses of 2 mg first alone on Day -1 and then co-administered with placebo matched to VX-973 on Day 27.
  Interventions: Drug: Placebo; Drug: Midazolam

INTERVENTIONS:
Drug: VX-973 — Suspension for oral administration.
  Arms: Part A: Single Ascending Dose; Part B: Multiple Ascending Dose
Drug: Placebo — Suspension for oral administration.
  Arms: Placebo Part A; Placebo Part B
Drug: Midazolam — Syrup for oral administration.
  Arms: Part B: Multiple Ascending Dose; Placebo Part B

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple doses of VX-973 in healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 32.0 kilogram per meter square (kg/m^2)
* A total body weight of more than (>) 50 kg
* Participants of non-childbearing potential
* Nonsmoker or ex-smoker for at least 3 months before screening

Key Exclusion Criteria:

* History of febrile illness or other acute illness that has not fully resolved within 14 days before the first dose of study drug
* Any condition possibly affecting drug absorption

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

PRIMARY OUTCOMES:
Part A: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 31
Part B: Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Day 1 up to Day 43

SECONDARY OUTCOMES:
Part A: Maximum Observed Plasma Concentration (Cmax) of VX-973 | From Day 1 up to Day 30
Part B: Maximum Observed Plasma Concentration (Cmax) of VX-973 | From Day 1 up to Day 43
Part A: Area Under the Concentration Versus Time Curve (AUC) of VX-973 | From Day 1 up to Day 30
Part B: Area Under the Concentration Versus Time Curve (AUC) of VX-973 | From Day 1 up to Day 43
Part B: Maximum Observed Plasma Concentration (Cmax) of Midazolam in the Absence and Presence of VX-973 | Days -1 and 27: Pre-dose up to 24 hours Post Midazolam dose
Part B: Area Under the Concentration Versus Time Curve (AUC) of Midazolam in the Absence and Presence of VX-973 | Days -1 and 27: Pre-dose up to 24 hours Post Midazolam dose

CONTACTS AND LOCATIONS:
Locations (1):
- PAREXEL International, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing